CLINICAL TRIAL: NCT04801914
Title: Influence of Percutaneous Biliary Drainage on the Change of Enzyme Activity of Matrix Metalloproteinases in the Serum of Patients With Malignant Obstructive Hyperbilirubinemia
Brief Title: Enzyme Activity of Matrix Metalloproteinases in the Serum of Patients With Malignant Obstructive Hyperbilirubinemia Before and After PTBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut za Rehabilitaciju Sokobanjska Beograd (Other)
Collaborators: Klinički centar Srbije (Unknown)
Responsible Party: Principal Investigator, Tamara Filipovic, Phd, Institut za Rehabilitaciju Sokobanjska Beograd
Other Study IDs: 717/11
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Matrix Metalloproteinase
Keywords: biliary drainage, matrix metalloproteinases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Matrix Metalloproteinases: Value of serum matrix metalloproteinase activity before and one month after PTBD
  Interventions: Procedure: Percutaneous biliary drainage

INTERVENTIONS:
Procedure: Percutaneous biliary drainage — Collection of peripheral blood samples before and one month after percutaneous biliary drainage performed for patients with malignant obstructive hyperbilirubinemia for further molecular biochemical analysis (measurement of serum matrix metalloproteinase activity).
  Other Names: Matrix Metalloproteinase serum activity measurement

SUMMARY:
The purpose of this study is to detect differences in the enzymatic activity of matrix metalloproteinases in patients with malignant obstructive hyperbilirubinemia before and after percutaneous biliary drainage.

DETAILED DESCRIPTION:
This study will be designed as a prospective cohort study involving the collection of peripheral blood samples before and one month after percutaneous biliary drainage for further molecular biochemical analysis (measurement of serum matrix metalloproteinase activity). Biochemical analyzes are preceded by the entry of data relevant to the research (demographic, anamnestic, clinical and biochemical).

ELIGIBILITY:
Inclusion Criteria:

pathological confirmation or imaging data confirming malignant disease causing bile duct obstruction, performance status 0-1

Exclusion Criteria:

terminally ill patients, performance status >2, hepatic decompensation, severe underlying cardiac or renal diseases and coagulation disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant obstructive hyperbilirubinemia admitted to hospital and referred to the interventional radiologist for percutaneous biliary drainage.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-03-11 (Estimated); Study Completion 2021-05-11 (Estimated)

PRIMARY OUTCOMES:
MMP-2 and MMP-9 serum activity | during intervention
  MMP serume activity will be measured by molecular biochemical analysis performed on peripheral blood samples taken before and one month after percutaneous biliary drainage

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gopcevic, Phd, Study Director — Institute for chemistry in medicine, Medical school, University of Belgrade
Locations (1):
- University Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No